CLINICAL TRIAL: NCT03152188
Title: Modulation of Gut-Brain Axis Using Fecal Transplant Capsules in Cirrhosis
Brief Title: Oral Fecal Transplant in Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: OpenBiome (Industry); Medical College of Wisconsin (Other); Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HM20009392; 1R21TR002024 (NIH)
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Hepatic Encephalopathy; Cirrhosis, Liver
Keywords: Hepatic Encephalopathy; Cirrhosis; Liver; Openbiome; FMT Capsule; Placebo
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Intervention Model Description: Placebo-controlled single-blind randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blind study in which subjects will not be aware whether they will be on placebo or FMT capsulres
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMT (Experimental): Fecal Microbiota Transplantation (FMT) capsules
  Interventions: Drug: FMT
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FMT — Fifteen FMT Openbiome capsules administered at the same time
  Arms: FMT
Other: Placebo — Fifteen placebo capsules administered at the same time
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of oral fecal transplant in patients with cirrhosis and hepatic encephalopathy

DETAILED DESCRIPTION:
Hepatic encephalopathy affects 30-45% of patients with cirrhosis and adversely affects survival in these patients. The mainstay of treatment for hepatic encephalopathy (HE) has long been the manipulation of the gut microbiota through antibiotics, prebiotics or probiotics. The current first and second line therapies for HE in the US are lactulose and rifaximin respectively that uniquely act within the confines of the gut lumen with encouraging clinical results. However there is a subset of patients with HE that continues to recur despite being on both treatments. This patient group is at a higher risk of poor outcomes because HE has now been removed from liver transplant priority and multiple episodes of HE can result in cumulative brain injury which may be irreversible. Therefore the prevention of recurrent HE is an important therapeutic goal.

The study team's research and other reports have shown that patients with HE and cirrhosis are more likely to have overgrowth of potentially pathogenic bacterial taxa such as Enterobacteriaceae and reduction of autochthonous species such as Lachnospiraceae and Ruminococcaceae in the stool and the colonic mucosa. This has been linked to poor performance on cognitive tests that are a hallmark of HE and with increased systemic inflammation in these patients.

Therefore a gut-based therapeutic option that can potentially improve the recurrence rate and the overall prognosis is needed. Fecal transplant has been shown to be effective in conditions with predominant gut-bacterial overgrowth or alteration such as recurrent Clostridium difficile and inflammatory bowel disease. Safe protocols have been developed across the world and studies are being performed in the US under FDA-monitored INDs. Limitations to performing fecal transplant include identifying and screening appropriate donors, which is time consuming and costly, with the cost typically falling to the patient or donor as the required screening is generally not covered by insurance. For this reason, the study team is particularly interested in working with Openbiome and have obtained their collaboration towards performing this Fecal Microbiota Transplantation (FMT) by cross-referencing of their drug master file.

The preliminary data suggest that a one-time administration of an FMT-enema using a rationally-selected donor via Openbiome is safe in patients with cirrhosis and recurrent HE. However, given the small bowel overgrowth and the predominantly small bowel location for bacterial translocation in cirrhosis, which is out of the reach of an enema, an upper GI route for FMT needs to be explored. The FMT capsule by Openbiome acts on the small and large intestine and is available for C.difficile. It is potentially more acceptable to patients for repeated administrations and in cirrhosis has the advantage of acting on the small bowel in addition to the large bowel. The study will use a donor specifically selected from the Openbiome pool whose microbial profile best fulfils the microbiota deficits related to beneficial bacteria in HE patients, utilizing a "Precision Microbiome" approach.

ELIGIBILITY:
Inclusion Criteria:

* 21-75 years of age
* Cirrhosis diagnosed by either of the following in a patient with chronic liver disease (a) Liver Biopsy (b) Radiologic evidence of varices, cirrhosis or portal hypertension (c) Laboratory evidence of platelet count <100,000 or AST/ALT ratio>1 (d) Endoscopic evidence of varices or portal gastropathy
* At least two HE episodes, one within the last year but not within the last month (patient can be on lactulose and rifaximin)
* Able to give written, informed consent (mini-mental status exam>25 at the time of consenting)

Exclusion Criteria:

Disease-related: (1) MELD score>17 (2) WBC count<1000 (3) TIPS, non-elective hospitalization or HE within last month (4) on dialysis (5) known untreated, in-situ luminal GI cancers (6) chronic intrinsic GI diseases (ulcerative colitis, Crohn's disease or microscopic colitis, eosinophilic gastroenteritis and celiac disease) Endoscopy-related: (1) Platelet count<50,000 (2) adverse reactions to sedation (3) lack of driver or other contra-indications Safety-related: (1) Dysphagia (2) History of aspiration, gastroparesis, intestinal obstruction (3) Ongoing absorbable antibiotic use (4) Severe anaphylactic food allergy (5) allergy to ingredients Generally Recognized As Safe in the G3 capsules (glycerol, sodium chloride, hypromellose, gellan gum, titanium dioxide, theobroma oil) (6) Adverse event attributable to prior FMT (7) ASA Class IV or V (8) Pregnant or nursing patients (9) acute illness or fever on the day of planned FMT

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Serious Adverse events related to FMT | 5 months
  Safety

SECONDARY OUTCOMES:
Frequency, severity and relatedness of solicited and unsolicited AEs | 5 months
  Safety
Occurrence of new potentially transmitted infections in the FMT group | 5 months
  Safety
Occurrence of new onset or significant worsening of chronic medical conditions post-FMT | 5 months
  Safety
changes in microbiota composition of the stool, duodenal and sigmoid colonic mucosa after oral FMT compared to pre-FMT baseline and donor compared to placebo post-FMT | 30 days
  Mechanism
mucosal defenses by studying antimicrobial peptides, inflammatory cytokine expression and barrier protein expression compared to pre-FMT baseline and compared to placebo | 30 days
  Mechanism
cognitive function after oral FMT compared to pre-FMT baseline and compared to placebo | 30 days
  Mechanism

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan Bajaj, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Bajaj JS, Salzman N, Acharya C, Takei H, Kakiyama G, Fagan A, White MB, Gavis EA, Holtz ML, Hayward M, Nittono H, Hylemon PB, Cox IJ, Williams R, Taylor-Robinson SD, Sterling RK, Matherly SC, Fuchs M, Lee H, Puri P, Stravitz RT, Sanyal AJ, Ajayi L, Le Guennec A, Atkinson RA, Siddiqui MS, Luketic V, Pandak WM, Sikaroodi M, Gillevet PM. Microbial functional change is linked with clinical outcomes after capsular fecal transplant in cirrhosis. JCI Insight. 2019 Dec 19;4(24):e133410. doi: 10.1172/jci.insight.133410. PMID 31751317
- [Derived] Bajaj JS, Salzman NH, Acharya C, Sterling RK, White MB, Gavis EA, Fagan A, Hayward M, Holtz ML, Matherly S, Lee H, Osman M, Siddiqui MS, Fuchs M, Puri P, Sikaroodi M, Gillevet PM. Fecal Microbial Transplant Capsules Are Safe in Hepatic Encephalopathy: A Phase 1, Randomized, Placebo-Controlled Trial. Hepatology. 2019 Nov;70(5):1690-1703. doi: 10.1002/hep.30690. Epub 2019 Jun 18. PMID 31038755